CLINICAL TRIAL: NCT02264639
Title: An Open Label, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of APL-2 as an Add-On to Standard of Care in Subjects With Paroxysmal Nocturnal Hemoglobinuria (PNH).
Brief Title: A Phase I Study to Assess the Safety of Pegcetacoplan (APL-2) as an Add-On to Standard of Care in Subjects With PNH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APL-CP0514
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: PNH; Paroxysmal Nocturnal Hemoglobinuria; Complement inhibitor; Anemia; Hemoglobinuria; hematologic diseases; extravascular hemolysis (EVH); intravascular hemolysis (IVH); C3 inhibitor
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Anemia; Hemoglobinuria; Hematologic Diseases; Hemolysis | interventions — pegcetacoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): First Dose 25mg, Repeated Dose 5 mg/day
  Interventions: Drug: Pegcetacoplan
- Cohort 2 (Experimental): First Dose 50 mg, Repeated Dose 30 mg/day
  Interventions: Drug: Pegcetacoplan
- Cohort 3 (Experimental): Repeated Dose 180 mg/day
  Interventions: Drug: Pegcetacoplan
- Cohort 4 (Experimental): Repeated Dose 270 mg/day
  Interventions: Drug: Pegcetacoplan

INTERVENTIONS:
Drug: Pegcetacoplan — Complement (C3) Inhibitor
  Other Names: APL-2

SUMMARY:
This study will be the initial exploration of pegcetacoplan in patients with PNH. The assessments of the safety, tolerability, PK, and PD following administration of single and multiples doses of pegcetacoplan will guide decisions to further develop the drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* At least 18 years of age
* Weigh >55 kg
* Diagnosed with PNH
* On treatment with eculizumab (Soliris®) for at least 3 months
* Hb < 10 g/dL at screening OR have received at least one transfusion within 12 months prior to screening
* Platelet count of >30,000/mm3
* Absolute neutrophil count > 500/mm3
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test at screening and must agree to use protocol defined methods of contraception for the duration of the study (see below)
* Males with female partners of child bearing potential must agree to use protocol defined methods of contraception (see below) and agree to refrain from donating sperm for the duration of the study
* Willing and able to give informed consent

Exclusion Criteria:

* Active bacterial infection
* Known infection with hepatitis B, C or HIV
* Hereditary complement deficiency
* History of bone marrow transplantation
* Participation in any other investigational drug trial or exposure to other investigational agent, device or procedure within 30 days
* Evidence of QTcF prolongation defined as > 450 ms for males and > 470 ms for females at screening
* Creatinine clearance (CrCl) < 50 mL/min (Cockcroft-Gault formula) at screening
* Breast-feeding women
* History of meningococcal disease
* No vaccination against N. meningitidis types A, C, W, Y and B (administered as two separate vaccinations), Pneumococcal conjugate vaccine or Pneumococcal polysaccharide vaccine 23 (PCV13 or PPSV23, respectively) and Haemophilus influenzae Type B (Hib) vaccination within 2 years prior to Day 1 (Visit 2) dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Grossi, MD, PhD, Study Director — Apellis Pharmaceuticals, Inc.
Locations (7):
- United States (7):
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - Lakes Research, Miami Lakes, Florida
  - University of Lousiville, Louisville, Kentucky
  - John Hopkins Hospital, Baltimore, Maryland
  - Cure 4 The Kids Foundation, Las Vegas, Nevada
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Paroxysmal nocturnal hemoglobinuria (PNH) subjects who were still anemic during treatment with eculizumab (Soliris®) were enrolled in this Phase 1, open-label, single- and multiple-ascending dose study to receive treatment with pegcetacoplan (APL-2) as an add-on to standard of care treatment. The study was conducted at 7 sites in the United States.
Pre-assignment Details: Subjects could participate in more than 1 cohort. Overall, 9 unique subjects were evaluated in 4 cohorts, with some subjects participating in >1 cohort. Single-dose phase: 4 unique subjects evaluated (2 each in Cohorts 1 and 2). Multiple-dose phase: 8 unique subjects evaluated, comprising 3 subjects who also participated in single-dose phase (1 in Cohort 1; 2 in Cohort 2) plus a further 5 unique subjects. Each cohort included a 30-day screening phase prior to treatment with pegcetacoplan.
Groups:
- Cohort 1 Single- and Multiple-dose Phase: Cohort 1 single-dose phase: Subjects received a single subcutaneous (SC) dose of 25 milligrams (mg) pegcetacoplan on Day 1.
  Cohort 1 multiple-dose phase: Following a waiting period of at least 28 days after single dosing, subjects received 5 mg/day SC dose of pegcetacoplan for 28 days (from Day 29 to Day 56).
- Cohort 2 Single- and Multiple-dose Phase: Cohort 2 single-dose phase: Subjects received a single SC dose of 50 mg pegcetacoplan on Day 1.
  Cohort 2 multiple-dose phase: Following a waiting period of at least 28 days after single dosing, subjects received 30 mg/day SC dose of pegcetacoplan for 28 days (from Day 29 to Day 56).
- Cohort 2 Single-dose Phase, Then Cohorts 2, 3, and 4 Multiple-dose Phase: Cohort 2 single-dose phase: Subjects received a single SC dose of 50 mg pegcetacoplan on Day 1.
  Cohort 2 multiple-dose phase: Following a waiting period of at least 28 days after single dosing, subjects received 30 mg/day SC dose of pegcetacoplan for 28 days (from Day 29 to Day 56).
  Cohort 3 multiple-dose phase: Subjects received 180 mg/day SC dose of pegcetacoplan for 28 days (from Day 1 to Day 28).
  Cohort 4 multiple-dose phase: Subjects received 270 mg/day SC doses of pegcetacoplan for up to 729 days (from Day 1 up to Day 729). The treatment period consisted of the following:
  * Part 1: Subjects received daily doses of pegcetacoplan for 28 days.
  * Part 2A: On Day 29, subjects who demonstrated clinical benefit from the treatment were automatically entered into Part 2A and continued to receive daily doses of pegcetacoplan until Day 84.
  * Part 2B: If there was ongoing evidence of clinical benefit, subjects who completed Part 2A could enter Part 2B and continue to receive daily doses of pegcetacoplan until Day 364.
  * Part 2C: If there was ongoing evidence of clinical benefit, subjects who completed Part 2B could enter Part 2C and continue to receive daily doses of pegcetacoplan until Day 729.
  After Day 28 (Part 1), individual subject dose escalation up to a dose of 360 mg/day could occur in subjects who had a sub-optimal hematological response but acceptable tolerability.
- Cohorts 3 and 4 Multiple-dose Phase: Cohort 3 multiple-dose phase: Subjects received 180 mg/day SC dose of pegcetacoplan for 28 days (from Day 1 to Day 28).
  Cohort 4 multiple-dose phase: Subjects received 270 mg/day SC doses of pegcetacoplan for up to 729 days (from Day 1 up to Day 729). The treatment period consisted of the following:
  * Part 1: Subjects received daily doses of pegcetacoplan for 28 days.
  * Part 2A: On Day 29, subjects who demonstrated clinical benefit from the treatment were automatically entered into Part 2A and continued to receive daily doses of pegcetacoplan until Day 84.
  * Part 2B: If there was ongoing evidence of clinical benefit, subjects who completed Part 2A could enter Part 2B and continue to receive daily doses of pegcetacoplan until Day 364.
  * Part 2C: If there was ongoing evidence of clinical benefit, subjects who completed Part 2B could enter Part 2C and continue to receive daily doses of pegcetacoplan until Day 729.
  After Day 28 (Part 1), individual subject dose escalation up to a dose of 360 mg/day could occur in subjects who had a sub-optimal hematological response but acceptable tolerability.
- Cohort 4 Multiple-dose Phase: Cohort 4 multiple-dose phase: Subjects received 270 mg/day SC doses of pegcetacoplan for up to 729 days (from Day 1 up to Day 729). The treatment period consisted of the following:
  * Part 1: Subjects received daily doses of pegcetacoplan for 28 days.
  * Part 2A: On Day 29, subjects who demonstrated clinical benefit from the treatment were automatically entered into Part 2A and continued to receive daily doses of pegcetacoplan until Day 84.
  * Part 2B: If there was ongoing evidence of clinical benefit, subjects who completed Part 2A could enter Part 2B and continue to receive daily doses of pegcetacoplan until Day 364.
  * Part 2C: If there was ongoing evidence of clinical benefit, subjects who completed Part 2B could enter Part 2C and continue to receive daily doses of pegcetacoplan until Day 729.
  After Day 28 (Part 1), individual subject dose escalation up to a dose of 360 mg/day could occur in subjects who had a sub-optimal hematological response but acceptable tolerability.
Period: Overall Study
Arm/Group | Cohort 1 Single- and Multiple-dose Phase | Cohort 2 Single- and Multiple-dose Phase | Cohort 2 Single-dose Phase, Then Cohorts 2, 3, and 4 Multiple-dose Phase | Cohorts 3 and 4 Multiple-dose Phase | Cohort 4 Multiple-dose Phase
Started | 2 (Subjects in this arm participated in Cohort 1 only.) | 1 (Subject in this arm participated in Cohort 2 only.) | 1 (Subject in this arm participated in Cohorts 2, 3 and 4.) | 1 (Subject in this arm participated in Cohorts 3 and 4; single-dose phase was not applicable.) | 4 (Subjects in this arm participated in Cohort 4 only; single-dose phase was not applicable.)
Completed (Completed the study (with reference to the last cohort in which a subject participated).) | 0 | 1 | 0 | 1 | 3
Not Completed | 2 | 0 | 1 | 0 | 1
Not completed — Death (after completing single-dose phase) | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by subject (during multiple-dose phase) | 1 | 0 | 0 | 0 | 0
Not completed — Pregnancy (during multiple-dose phase) | 0 | 0 | 1 | 0 | 0
Not completed — Major Intercurrent Illness (during multiple-dose phase) | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all enrolled subjects who received at least 1 dose of study drug. Total unique participants = 9. Subjects could participate in more than 1 cohort. 1 subject participated in Cohorts 2, 3 and 4, and 1 subject participated in Cohorts 3 and 4.
Groups:
- Cohort 1 Single- and Multiple-dose Phase: Cohort 1 single-dose phase: Subjects received a single SC dose of 25 mg pegcetacoplan on Day 1.
  Cohort 1 multiple-dose phase: Following a waiting period of at least 28 days after single dosing, subjects received 5 mg/day SC dose of pegcetacoplan for 28 days (from Day 29 to Day 56).
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Single- and Multiple-dose Phase | Cohort 2 Single- and Multiple-dose Phase | Cohort 2 Single-dose Phase, Then Cohorts 2, 3, and 4 Multiple-dose Phase | Cohorts 3 and 4 Multiple-dose Phase | Cohort 4 Multiple-dose Phase | Total
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 1 | 4 | 8
  >=65 years | 1 | 0 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 1 | 4 | 8
  Male | 0 | 1 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 1 | 1 | 0 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1
  White | 2 | 1 | 1 | 1 | 3 | 8
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 1 | 1 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs), Including by Severity, During Single-dose Phase
Description: TEAEs were defined as AEs that developed or worsened after first dose of study drug (Day 1), and up to 30 days after last dose of study drug. The Investigator assessed AEs for severity and relatedness to study drug. AEs were graded according to the Common Terminology Criteria for Adverse Events (CTCAE, v4.03) based on: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death related to AE.
Time Frame: From single dose of study drug (Day 1) up to 30 days
Population: The safety population included all enrolled subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 Single-dose Phase: Subjects received a single SC dose of 25 mg pegcetacoplan on Day 1.
- Cohort 2 Single-dose Phase: Subjects received a single SC dose of 50 mg pegcetacoplan on Day 1.
Arm/Group | Cohort 1 Single-dose Phase | Cohort 2 Single-dose Phase
Number analyzed (Participants) | 2 | 2
Participants
  Any TEAE | 1 | 2
  TEAE at least possibly related to study drug | 0 | 1
  Serious TEAE | 0 | 0
  TEAE leading to study drug discontinuation | 0 | 0
  TEAE leading to death | 0 | 0
  Maximum severity of all TEAEs: mild | 0 | 1
  Maximum severity of all TEAEs: moderate | 1 | 1
  Maximum severity of all TEAEs: severe | 0 | 0

2. Primary Outcome: Number of Subjects With TEAEs, Including by Severity, During Multiple-dose Phase
Description: TEAEs were defined as AEs that developed or worsened after first dose of study drug (Day 1), and up to 30 days after last dose of study drug. The Investigator assessed AEs for severity and relatedness to study drug. AEs were graded according to CTCAE, v4.03 based on: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death related to AE.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (Cohorts 1-3: up to 58 days; Cohort 4: up to 759 days).
Population: The safety population included all enrolled subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 Multiple-dose Phase: Subjects received 5 mg/day SC dose of pegcetacoplan for 28 days (from Day 29 to Day 56).
- Cohort 2 Multiple-dose Phase: Subjects received 30 mg/day SC dose of pegcetacoplan for 28 days (from Day 29 to Day 56).
- Cohort 3 Multiple-dose Phase: Subjects received 180 mg/day SC dose of pegcetacoplan for 28 days (from Day 1 to Day 28).
- Cohort 4 Multiple-dose Phase: Subjects received 270 mg/day SC dose of pegcetacoplan for up to 729 days (from Day 1 up to Day 729).
  After Day 28, individual subject dose escalation up to a dose of 360 mg/day could occur in subjects who had a sub-optimal hematological response but acceptable tolerability.
Arm/Group | Cohort 1 Multiple-dose Phase | Cohort 2 Multiple-dose Phase | Cohort 3 Multiple-dose Phase | Cohort 4 Multiple-dose Phase
Number analyzed (Participants) | 1 | 2 | 2 | 6
Participants
  Any TEAE | 1 | 2 | 1 | 6
  TEAE at least possibly related to study drug | 0 | 1 | 1 | 4
  Serious TEAE | 0 | 0 | 0 | 2
  TEAE leading to study drug discontinuation | 1 | 0 | 0 | 0
  TEAE leading to death | 0 | 0 | 0 | 0
  Maximum severity of all TEAEs: mild | 0 | 0 | 1 | 0
  Maximum severity of all TEAEs: moderate | 0 | 2 | 0 | 2
  Maximum severity of all TEAEs: severe | 1 | 0 | 0 | 4
  Maximum severity of all TEAEs: life-threatening | 0 | 0 | 0 | 0

3. Primary Outcome: Area Under the Curve (AUC) From Time 0 to the Last Measurable Concentration (AUC0-t) Over the Multiple Dosing Phase for Cohort 4
Description: Assessment of AUC0-t of pegcetacoplan over the multiple dosing phase, estimated using a non-compartmental approach and calculated by the linear-log trapezoidal method. Pegcetacoplan pharmacokinetic (PK) parameters were summarized for Cohort 4 only.
Time Frame: Blood samples for PK assessment were collected pre-dose and 4 hours post dose on Day 1 and pre-dose (trough) on Day 2 and up to Day 785.
Population: The PK population was defined as all subjects in the safety population who had at least 1 PK sample drawn with a measurable serum concentration. Results were reported for Cohort 4 only. Due to the small sample size in Cohorts 1 through 3, summaries for continuous data using descriptive statistics were not performed.
Measure: Mean (Standard Deviation); unit: micrograms*hour/milliliter (μg*hour/mL)
Arm/Group | Cohort 4 Multiple-dose Phase
Number analyzed (Participants) | 6
micrograms*hour/milliliter (μg*hour/mL) | 6,500,000 (3,990,000)

4. Primary Outcome: Maximum Pre-dose Serum Concentration (Ctrough,Max) Over the Multiple Dosing Phase for Cohort 4
Description: Assessment of Ctrough,max of pegcetacoplan over the multiple dosing phase, estimated using a non-compartmental approach. Pegcetacoplan PK parameters were summarized for Cohort 4 only. Ctrough,max was calculated for both 270 mg/day and 360 mg/day where subjects received both doses. Note: 1 subject in Cohort 4 who was receiving 360 mg/day was granted Sponsor and institutional review board approval to increase the dose further to the equivalent of 440 mg/day and Ctrough,max is also reported for this dose.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cohort 4 Multiple-dose Phase
Number analyzed (Participants) | 6
μg/mL
  270 mg Dose | 627 (207)
  360 mg Dose: number analyzed (Participants) | 4
  360 mg Dose | 543 (192)
  440 mg Dose: number analyzed (Participants) | 1
  440 mg Dose | 624 (NA) — No standard deviation is presented since mean value is derived from a single subject.

ADVERSE EVENTS:
Time Frame: TEAE data is reported from first dose of study drug up to 30 days after last dose of study drug (Cohorts 1 and 2, single-dose phase: up to 30 days; Cohorts 1-3, multiple-dose phase: up to 58 days; Cohort 4, multiple-dose phase: up to 759 days).
Description: The safety population included all enrolled subjects who received at least 1 dose of study drug. The 4 cohorts of 12 subjects overall represents 9 unique participants. Subjects could participate in more than 1 cohort. The all-cause mortality table includes the death of 1 subject in Cohort 1, resulting from a serious AE which was not treatment-emergent.
Groups:
- Cohort 1 Multiple-dose Phase: Subjects received pegcetacoplan 5 mg/day as SC dose for 28 days (from Day 29 to Day 56).
- Cohort 2 Multiple-dose Phase: Subjects received pegcetacoplan 30 mg/day as SC dose for 28 days (from Day 29 to Day 56).
- Cohort 3 Multiple-dose Phase: Subjects received pegcetacoplan 180 mg/day as SC dose for 28 days (from Day 1 to Day 28).
- Cohort 4 Multiple-dose Phase: Subjects received pegcetacoplan 270 mg/day as SC dose for up to 729 days (from Day 1 up to Day 729).
  After Day 28, individual subject dose escalation up to a dose of 360 mg/day could occur in subjects who had a sub-optimal hematological response but acceptable tolerability.
Arm/Group | Cohort 1 Single-dose Phase | Cohort 2 Single-dose Phase | Cohort 1 Multiple-dose Phase | Cohort 2 Multiple-dose Phase | Cohort 3 Multiple-dose Phase | Cohort 4 Multiple-dose Phase
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/2 | 0/1 | 0/2 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/1 | 0/2 | 0/2 | 2/6
Other Adverse Events (participants affected / at risk) | 1/2 | 2/2 | 1/1 | 2/2 | 1/2 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Single-dose Phase (N=2) | Cohort 2 Single-dose Phase (N=2) | Cohort 1 Multiple-dose Phase (N=1) | Cohort 2 Multiple-dose Phase (N=2) | Cohort 3 Multiple-dose Phase (N=2) | Cohort 4 Multiple-dose Phase (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Single-dose Phase (N=2) | Cohort 2 Single-dose Phase (N=2) | Cohort 1 Multiple-dose Phase (N=1) | Cohort 2 Multiple-dose Phase (N=2) | Cohort 3 Multiple-dose Phase (N=2) | Cohort 4 Multiple-dose Phase (N=6)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (5)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum ferritin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection-site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 4 (145)
Injection-site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (43)
Injection-site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (19)
Injection-site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (13)
Injection-site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (9)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8)
Injection-site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7)
Infusion-site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injection-site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection-site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection-site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection-site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (9)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin B12 decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (11)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diplopia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT02264639/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT02264639/SAP_001.pdf